CLINICAL TRIAL: NCT03443180
Title: Gluten and Amylase Trypsin Inhibitors (ATI) as Nutritional Contributors to Type 1 Diabetes Susceptibility
Brief Title: Gluten and Amylase Trypsin Inhibitors (ATI) Free Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Susanne Cabrera, Principal Investigator, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1138159
Record Dates: First submitted 2018-01-31; First posted 2018-02-23 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Type1diabetes
Keywords: Siblings
MeSH Terms: interventions — Glutens

STUDY DESIGN:
Intervention Model Description: All subjects will receive a dietary intervention. They will be instructed and asked to follow a diet free of gluten and the protein amylase trypsin inhibitors (ATI), which is frequently found in gluten-containing foods, for four weeks. They will then be asked to resume their normal diet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dietary intervention (Other): Participants will be asked to remove food containing gluten and ATI from their diets for 4 weeks.
  Interventions: Other: Gluten and Amylase Trypsin Inhibitors (ATI)-free diet

INTERVENTIONS:
Other: Gluten and Amylase Trypsin Inhibitors (ATI)-free diet — Participants will be asked to avoid foods containing gluten and ATI (a similar protein found in grains) for 4 weeks.

SUMMARY:
Siblings of those with type 1 diabetes are at an increased risk of developing the disease themselves. Through prior research, the investigators have found that siblings as well as those with type 1 diabetes have a general level of inflammation in the body. The investigators are examining the role that diet plays in this level of inflammation by asking siblings of children with type 1 diabetes to go on a gluten and Amylase Trypsin Inhibitors (ATI)-free diet for 4 weeks. Blood and stool samples will be measured before the diet, after the diet is completed and again 4 weeks after participants resume their normal diet.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 2-23 years of age
2. Full-sibling of an individual with a clinical diagnosis of type 1 diabetes
3. Treatment naïve of any immunomodulatory agent

Exclusion Criteria:

1. Abnormal HbA1c, defined as ≥ 6%
2. Previous or current use of a gluten-free diet
3. Current diagnosis of celiac disease
4. An elevated tissue transglutaminase IgA level (> 10 units/mL)
5. Chronic (≥ 3 months duration) gastrointestinal disease or presence of gastrointestinal symptoms within the prior 6 weeks (e.g., abdominal pain, worsening constipation, diarrhea, or recurrent nausea +/- vomiting)
6. Chronic inflammatory or autoimmune disease with the exception of well-controlled hypothyroidism or intermittent or mild persistent asthma not requiring the use of daily inhaled steroids
7. Use of any medications that affect glucose metabolism (e.g., metformin) or the immune system (e.g., use of any glucocorticoids (inhaled, intranasal, oral, intravenous) within the previous 3 months)
8. Use of any medications that could affect intestinal microbiota within the previous 3 months (e.g., antibiotics, prebiotics, or probiotics)
9. Any condition that, in the investigator's opinion, may compromise study participation or may confound the interpretation of the study results

Ages: 2 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
Change in the plasma-induced transcriptional assay | 2 years (study duration)
  Investigators will measure the participants overall immune inflammation and regulation by a plasma-induced transcriptional bioassay. The change in this bioassay will be determined for each subject and the entire group both before and after the dietary intervention. This bioassay informs the investigators of which genes may be positively or negatively impacted by this dietary change and whether the removal of gluten and amylase trypsin inhibitors (ATI) affects a participant's immune state.

SECONDARY OUTCOMES:
Stool microbial composition | 2 years (study duration)
  Stool samples will be collected both before and after the dietary intervention to determine if the removal of gluten and amylase trypsin inhibitors (ATI) from the diet affects the composition and density of the stool microbiota
Plasma microbial antigen detection | 2 years (study duration)
  Microbial antigen levels in the plasma of participants will be assayed both before and after the dietary intervention. Systemic microbial antigens are a marker of intestinal permeability so this measure will tell the investigators if the removal of gluten and amylase trypsin inhibitors (ATI) affects the degree of intestinal permeability/leakiness.
Leukocyte analyses | 2 years (study duration)
  The degree of responsiveness of participants leukocytes to stimulation with gluten and amylase trypsin inhibitors (ATI) will be measured in vitro both before and after the dietary intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided